CLINICAL TRIAL: NCT00312754
Title: A Phase IV, One-arm, Open-label, Multicenter Study Evaluating Effect of Treatment Change to Atazanavir/Ritonavir on Brachial Endothelial Function of HIV Infected Patient Receiving Function in HIV Infected Patient Receiving Potent Antiretroviral Combination Therapy
Brief Title: A Phase IV Study of BMS-232632 in HIV+ Patients With Metabolic Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI424-108; Amazone
Record Dates: First submitted 2005-11-14; First posted 2006-04-11 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate

INTERVENTIONS:
Drug: Atazanavir

SUMMARY:
The purpose of this clinical research study is to learn if BMS-232632 administered as Atazanavir/ritonavir (ATV/RTV) is superior to an anti-retroviral regimen including Lopinavir/ritonavir (LPV/RTV), as assessed by an increased brachial artery flow-mediated vasodilatation (FMD), in HIV-infected patients. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

- Documented Metabolic Syndrome by at least 3 of the following parameters:

* Abdominal obesity, assessed by waist circumference (for men >103 cm, for women >88 cm).
* Triglycerides > 150 mg/dl.
* HDL cholestrol (for men <40 mg/dl, for women <50 mg/dl).
* Blood pressure > or equal to 130/85 mm Hg.
* Fasting serum glucose > or equal to 110 mg/dl.
* HIV RNA < 50 copies/mL.
* IP within 3 months prior to selection.

Exclusion Criteria:

-Treated Metabolic Syndrom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2005-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To demonstrate a significant increase in brachial artery FMD after a 24-week ATV/RTV treatment period.

SECONDARY OUTCOMES:
The change in FMD from ref. value after a 12-wk ATV/RTV treatment period.
The proportion of pts w/ virologic rebound after a 24-wk ATV/RTV treatment period.
The proportion of pts w/ metabolic syndrome after a 24-wk ATV/RTV treament period.-

CONTACTS AND LOCATIONS:
Overall Officials: Yacia Bennai, MD, Study Director — 00 33 1 58 83 63 84
Locations (3):
- France (3):
  - Local Institution, Bobigny
  - Local Institution, Le Kremlin-Bicêtre
  - Local Institution, Paris